CLINICAL TRIAL: NCT01460693
Title: A Phase III, Prospective Randomised Comparison of Imatinib (STI571, Glivec/Gleevec) 400mg Daily Versus Dasatinib 100mg in Patients With Newly-diagnosed Chronic Phase Chronic Myeloid Leukaemia
Brief Title: Comparison of Imatinib Versus Dasatinib in Patients With Newly-diagnosed Chronic Phase Chronic Myeloid Leukaemia
Acronym: SPIRIT2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Newcastle University (Other)
Collaborators: Newcastle-upon-Tyne Hospitals NHS Trust (Other); Bristol-Myers Squibb (Industry); Institute of Cancer Research, United Kingdom (Other); Hammersmith Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4443; 2007-006185-15 (EudraCT Number); ISRCTN54923521 (Other: ISRCTN)
Record Dates: First submitted 2010-10-01; First posted 2011-10-27 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Myeloid Leukemia, Chronic, Chronic Phase
Keywords: Leukemia; Myeloid; Chronic; Chronic-Phase; CML
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase; Leukemia; Bronchiolitis Obliterans Syndrome | interventions — Imatinib Mesylate; Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A - Imatinib (Active Comparator): Imatinib 400mg daily
  Interventions: Drug: Imatinib
- Arm B - Dasatinib (Experimental): Dasatinib 100mg daily
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Imatinib — Oral Imatinib 100mg daily
  Other Names: Gleevec/Gleevic
  Arms: Arm A - Imatinib
Drug: Dasatinib — Oral Dasatinib 100mg daily
  Other Names: Sprycel
  Arms: Arm B - Dasatinib

SUMMARY:
Imatinib 400mg daily is the current NICE-approved standard treatment for newly diagnosed Chronic Myeloid Leukaemia (CML). 5 yr follow up of CML patients treated in this way indicates an 89% probability of progression-free survival. Imatinib is not tolerated or effective in some patients however, and a proportion of patients become resistant to the drug. SPIRIT 2 study aims to establish whether a new drug, dasatinib, is superior to imatinib in terms of event free survival and therefore will be an effective first-line therapy for newly-diagnosed CML patients. This study will also provide crucial long-term survival, quality of life and health economic data to assist health care providers and managers to determine the most cost-effective drug therapy for CML.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 18 years or over.
2. Patients must have all of the following:

   * be enrolled within 3 months of initial diagnosis of CML-CP (date of initial diagnosis is the date of first cytogenetic analysis)
   * cytogenetic confirmation of the Philadelphia chromosome or variants of (9;22) translocations
   * patients may have secondary chromosomal abnormalities in addition to the Philadelphia chromosome.
   * < 15% blasts in peripheral blood and bone marrow;
   * < 30% blasts plus promyelocytes in peripheral blood and bone marrow;
   * < 20% basophils in peripheral blood,
   * 100 x 109/L platelets or greater
   * no evidence of extramedullary leukaemic involvement, with the exception of the hepatosplenomegaly.
3. Written voluntary informed consent.

Exclusion Criteria:

1. Patients with Ph-negative, BCR-ABL-positive, disease are NOT eligible for the study.
2. Any prior treatment for CML with: any tyrosine kinase inhibitor (eg imatinib, dasatinib); busulphan; interferon-alpha; homoharringtonine; cytosine arabinoside; any other investigational agents (hydroxycarbamide and anagrelide are the only drugs permitted). NB patients will be ineligible for the study if they have received ANY prior therapy with interferon-alpha or imatinib. NO exceptions.
3. Patients who received prior chemotherapy, including regimens used in peripheral blood progenitor cells (PBPCs) mobilisation for haematopoietic progenitor-cell transplantation. (It is allowable to collect unmobilised PBPCs at diagnosis.)
4. Patient who have had any form of prior haemopoietic stem cell transplant, either autograft or allograft.
5. Patients with an ECOG Performance Status Score of 2 or less.
6. Patients with serum bilirubin, SGOT/AST, SGPT/ALT, or creatinine concentrations > 2.0 x the institutional upper limit of the normal range (IULN).
7. Patients with International normalized ratio (INR) or partial thromboplastin time (PTT) > 1.5 x IULN, with the exception of patients on treatment with oral anticoagulants.
8. Patients with uncontrolled medical disease such as diabetes mellitus, thyroid dysfunction, neuropsychiatric disorders, infection, angina, or Grade 3/4 cardiac problems as defined by the New York Heart Association Criteria.
9. Patients with known positivity for human immunodeficiency virus (HIV); baseline testing for HIV is not required.
10. Patients who have undergone major surgery within 4 weeks of Study Day 1, or who have not recovered from prior major surgery.
11. Patients who are:

    * pregnant,
    * breast feeding,
    * of childbearing potential without a negative pregnancy test prior to Study Day 1, and
    * male or female of childbearing potential unwilling to use barrier contraceptive precautions throughout the trial (postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential).
12. Patients with a history of another malignancy either currently or within the past five years, with the exception of basal cell skin carcinoma or cervical carcinoma in situ.
13. Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 814 (Actual)
Dates: Start 2008-08; Primary Completion 2018-03-07 (Actual); Study Completion 2018-03-07 (Actual)

PRIMARY OUTCOMES:
5-year event free survival | ongoing throughout study (5 years)
  To compare 5-year event free survival between the 2 treatment arms. The study aim is to show superiority of the dasatinib arm over the imatinib 400mg arm.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen G O'Brien, MD, Principal Investigator — Newcastle University; Richard E Clark, MD, Principal Investigator — Royal Liverpool University Hospital; Jane Apperley, MD, Principal Investigator — Imperial College London
Locations (1):
- Freeman Hospital, Newcastle upon Tyne, United Kingdom

REFERENCES:
- [Derived] Neelakantan P, Gerrard G, Lucas C, Milojkovic D, May P, Wang L, Paliompeis C, Bua M, Reid A, Rezvani K, O'Brien S, Clark R, Goldman J, Marin D. Combining BCR-ABL1 transcript levels at 3 and 6 months in chronic myeloid leukemia: implications for early intervention strategies. Blood. 2013 Apr 4;121(14):2739-42. doi: 10.1182/blood-2012-11-466037. Epub 2013 Feb 4. PMID 23380743
- [Derived] Marin D, Hedgley C, Clark RE, Apperley J, Foroni L, Milojkovic D, Pocock C, Goldman JM, O'Brien S. Predictive value of early molecular response in patients with chronic myeloid leukemia treated with first-line dasatinib. Blood. 2012 Jul 12;120(2):291-4. doi: 10.1182/blood-2012-01-407486. Epub 2012 May 29. PMID 22645182
- See also: Study website — http://www.spirit-cml.org